CLINICAL TRIAL: NCT00324246
Title: Feasibility Study of the NEW NORMA-SENSE Indicator Strip and Vaginal Secretion Buffer Capacity Measurement - IN-VITRO Study.
Brief Title: Feasibility Study of the NEW NORMA-SENSE
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Collaborators: Lin Medical Center, Haifa (Other); Common Sense (Other)
Responsible Party: hadar kessary, common sense
Other Study IDs: F-7-28-1 CTIL; CMC 06014008
Record Dates: First submitted 2006-05-09; First posted 2006-05-10 (Estimated); Last update posted 2008-06-20 (Estimated); Status verified 2007-01

CONDITIONS: Vaginal Infection
Keywords: vaginal infection; color appearance; new developed indicator strips (NEW NORMA-SENSE); in-vitro; vaginal secretion; elevated pH
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Vaginal secretions.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
* In-vitro study
* Collect data regarding the color appearance on the new developed indicator strips (NEW NORMA-SENSE), in contact with vaginal secretion with elevated pH
* Measure the buffering capacity of vaginal secretion from non-symptomatic and symptomatic subjects
* Detect these indicator strips' performance, in contact with urine

DETAILED DESCRIPTION:
This in-vitro study was designed to collect data regarding the color appearance on the new developed indicator strips (NEW NORMA-SENSE) when coming in contact, in-vitro, with vaginal secretion with elevated pH, and to measure the buffering capacity of vaginal secretion from non-symptomatic subjects and symptomatic subjects, and to detect these indicator strips' performance when come in contact with urine.

ELIGIBILITY:
Inclusion Criteria:

1. Women, aged between 18 and 45, with or without symptoms of vaginal infection.
2. Subjects are ready to sign the informed consent form.

Exclusion Criteria:

1. Subjects are unable or unwilling to cooperate with the study procedures.
2. Subjects are currently participating in another clinical study that may directly or indirectly affect the results of this study.
3. Subjects that suffer from vaginal bleeding or menstruate.
4. Subjects that have had sexual relations within the last 12 hours.
5. Subjects that applied local antiseptic, antibiotic or vaginal treatment within the last 3 days.
6. Subjects that applied vaginal douching within 12 hours prior to the visit at the clinic.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women, age between 18 years and 45 years with or without symptoms of vaginal infection.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2006-09; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Geva, MD, Principal Investigator — Women Health Care Center - Lin Medical Center, Haifa, Israel
Locations (1):
- Women Health Care Center - Lin Medical Center, Haifa, Israel